CLINICAL TRIAL: NCT04877574
Title: Effects of Analgesia Nociception Index (ANI)-Guided Intraoperative Analgesia on Postoperative Pain: a Randomized Controlled Study
Brief Title: ANI-guided Intraoperative Analgesia vs Conventional Intraoperative Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2104-033-1209
Record Dates: First submitted 2021-04-30; First posted 2021-05-07 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Postoperative Pain; Analgesia; Surgery
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ANI-guided intraoperative analgesia (Experimental): Intraoperative analgesia is performed by controlling the effect-site concentration of remifentanil to maintain 50-70 of ANI index.
  Interventions: Procedure: ANI-guided intraoperative analgesia
- Conventional intraoperative analgesia (Active Comparator): Intraoperative analgesia is performed by controlling the effect-site concentration of remifentanil at the discretion of attending anesthesiologists based on hemodynamic parameters.
  Interventions: Procedure: Conventional intraoperative analgesia

INTERVENTIONS:
Procedure: ANI-guided intraoperative analgesia — Intraoperative analgesia is performed by controlling the effect-site concentration of remifentanil to maintain 50-70 of ANI.
  Arms: ANI-guided intraoperative analgesia
Procedure: Conventional intraoperative analgesia — Intraoperative analgesia is performed by controlling the effect-site concentration of remifentanil at the discretion of attending anesthesiologists based on hemodynamic parameters.
  Arms: Conventional intraoperative analgesia

SUMMARY:
This study evaluates the effects of Analgesia Nociception Index (ANI)-guided intraoperative analgesia on postoperative pain in patients undergoing open gynecologic surgery.

DETAILED DESCRIPTION:
Postoperative pain is one of the most common postoperative complications and is significantly associated with patient's quality of recovery. Analgesia Nociception Index (ANI) is known to analyze the high frequency component of heart rate variability in relation to respiratory frequency, providing the objective information on the degree of pain. However, most previous studies conducted by using ANI were observational studies or small-sized randomized controlled studies. In the present study, the investigators aimed to evaluate the effects of ANI-guided intraoperative analgesia on moderate-to-severe postoperative pain by performing randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Elective open gynecological surgery
* American Society of Anaesthesiologists physical status classification 1-3

Exclusion Criteria:

* Laparoscopic surgery or robot-assisted surgery
* Patients who had analgesic agents, anti-psychotic agents, anticonvulsants which were related to chronic pain
* Patients who had hypersensitivity to analgesic agents or medications related anesthesia.
* Patients who were required to have mechanical ventilation after surgery
* Patients who had arrhythmia
* Patients who transferred to the surgical intensive care unit immediately after surgery
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
the incidence of moderate-to-severe postoperative pain | during 1 hour of stay in the postanesthesia care unit
  the incidence of moderate-to-severe postoperative pain is defined as a case in which pain with numeric rating scale (NRS) of 5 or more is reported during stays in the postanesthesia care unit. Pain assessment is performed two times during stays in the postanesthesia care unit.

SECONDARY OUTCOMES:
the amount of intraoperative remifentanil | intraoperative
  the amount of intraoperative remifentanil used during anesthesia
Quality of Recovery-15 (QoR-15) score | at postoperative 24 hour
  QoR-15 questionnaire is recorded by an investigator. QoR-15 questionnaire has minimum score of 0 and maximum score of 150, and higher score indicates the better quality of recovery.
the incidence of postoperative nausea and vomiting | at postoperative 1 hour, 24 hour, 72 hour
  the incidence of postoperative nausea and vomiting is recorded by an investigator
11-pointed NRS pain score | at postoperative 24 hour
  11-pointed NRS pain score is measured at both resting state and movement. 11-pointed NRS pain score has minimum score of 0 and maximum score of 10, and higher score indicates the higher severity of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No